CLINICAL TRIAL: NCT05449353
Title: Trauma-informed Cognitive Behavioural Therapy (TiCBT) to Aid Reintegration of Repentant Terrorists and Their Families in Nigeria: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tarela Ike (Other)
Collaborators: British International Studies Association (Unknown)
Responsible Party: Sponsor-Investigator, Tarela Ike, Dr, Teesside University
Organization: Teesside University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313a
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Trauma; Psychological
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-infomed Cognitive Behavioural Therapy (Experimental): Experimental (n=24 participants) will receive the TiCBT which consists of a total of 8-group integrated sessions lasting approximately 60 minutes per session every 3 days interval with 24 persons in the single group.
  Interventions: Behavioral: Trauma-informed Cognitive Behaviour Therapy (TiCBT)

INTERVENTIONS:
Behavioral: Trauma-informed Cognitive Behaviour Therapy (TiCBT) — Group: Experimental (n=24 participants) will receive the TiCBT which consists of a total of 8-group integrated sessions lasting approximately 60 minutes per session every 3 days interval with 24 persons in the single group.

SUMMARY:
The aim of the study is to describe the feasibility, cultural appropriateness, and acceptability of Trauma-informed Cognitive Behaviour Therapy (TiCBT) to promote community healing and encourage the reintegration of repentant terrorists and their families to avoid reoffending.

DETAILED DESCRIPTION:
The study will adopt a mixed-method single-arm experimental design. Approximately 24 participants will be recruited for the intervention. The Trauma-informed Cognitive Behaviour Therapy (TiCBT) is an 8-session intervention lasting approximately 1 hour each and designed to address trauma, dispel negative attitudes and encourage positive behaviour towards repentant terrorists. Measurement will be collected at baseline pre-intervention, end of intervention and three months post-intervention to determine its feasibility and effectiveness. Interviews will also be conducted post-intervention. Repeated-measures univariate analyses of variance (ANOVA) will be performed to examine differences between the pre- and post-intervention stages. Interviews will be analysed using thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* community members who are victims of Boko Haram terrorism and had previous experiences of trauma/depression,
* score five and above for the culturally-adapted Trauma Screening Questionnaire (Brewinn et al., 2002)
* aged 18+ years,
* able to give informed consent,
* speak English
* are residents or from areas within Nigeria including Maiduguri, Adamawa, and Plateau environs.

Exclusion Criteria:

* less than 18 or above 85 years
* unable to give consent
* clinically diagnosed with severe PTSD/suicidal ideations or undergoing treatment
* temporary or non-residents who are unlikely to be available for follow up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Trauma Screening Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in traumatic experience is being assessed
Patient Health Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in depression is being assessed
Attitude Towards Repentant Terrorists and their Reintegration Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in of attitude towards repentant terrorists is being assessed
brief Verona Service Satisfaction Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in service satisfaction is being assessed

IPD SHARING:
Plan to Share IPD: No